CLINICAL TRIAL: NCT02647814
Title: Salud al Día: Engaging Latino Parents in Pediatric Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gordon and Betty Moore Foundation (Other); emocha Mobile Health, Inc. (Other); Maryland Institute College of Art (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00075868
Record Dates: First submitted 2015-12-18; First posted 2016-01-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Primary Health Care
Keywords: Parent activation; Text-messages; LEP; Latino populations; pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salud al Día (Experimental): The participants in the intervention group will receive interactive text-messages with a link to support if needed for: clinic appointment reminders, follow-up on medicine and referral adherence, and illness care needs and use. Participants will additionally receive reminders for insurance renewal, food stamp applications, and health-promoting community events. Participants in this arm will complete a baseline survey when their infant is ≤ 2 months of age, a mid-point survey at 7-9 months, and a follow-up survey at by age 15 months.
  Interventions: Behavioral: Salud al Día
- Usual Care (No Intervention): The participants in the usual care group will receive the clinic's usual care in terms of receiving no text messages. Participants in this arm will complete a baseline survey when their infant is ≤ 2 months of age, a mid-point survey at 7-9 months, and a follow-up survey at by age 15 months.

INTERVENTIONS:
Behavioral: Salud al Día — A pilot randomized controlled trial comparing the effectiveness of a parent support intervention consisting of periodic text messages and educational support (video, collateral materials),and usual care on the healthcare engagement of LEP Latino parents during their child's first year and to examine its impact on healthcare utilization and primary care quality.
  Arms: Salud al Día

SUMMARY:
Objective: To conduct a pilot randomized controlled trial comparing the effectiveness of a parent support intervention consisting of periodic text messages and educational support (video, collateral materials),and usual care on the healthcare engagement of limited English proficient (LEP) Latino parents during participants' child's first year and to examine its impact on healthcare utilization and primary care quality.

DETAILED DESCRIPTION:
Lessons learned in organizational engagement reveal a critical need to increase healthcare engagement among LEP Latino parents. LEP Latina mothers who were founding members of Latino Family Advisory Board (LFAB) at the Johns Hopkins Bayview Medical Center identified the health system knowledge that enabled participants to more effectively use the healthcare system as one of the key benefits of board membership. The gains in knowledge, skills, and confidence demonstrated in the LFAB evaluation mirror qualitative evaluation findings of other ambulatory care advisory boards, and reflect the concept of patient activation. Patient activation, a component of individual patient engagement, is defined as the patient's willingness to manage their health and healthcare based on understanding one's role in the care process and having the knowledge, skills, and confidence to do so. Interventions focused on increasing activation, using both in-person and mHealth support, have demonstrated efficacy and have led to improvement in health and healthcare quality. mHealth-based interventions have the ability to reach larger populations at lower cost, with the potential for increased tailoring and interactivity, especially as the use of cellular phones becomes nearly universal, even among low-income populations. For example, Text4baby, a perinatal health education program delivered through passive educational text messages, has demonstrated success at reaching low-income Spanish-speaking parents with positive user assessments.

A recent study of parent healthcare activation among low-income parents (conducted by PI: DeCamp) demonstrated that parent activation among parents whose preferred healthcare language was Spanish was significantly lower than that of parents whose preferred healthcare language was English. These findings further support targeting increasing the healthcare engagement of LEP Latino parents.

This novel intervention will integrate mobile health (mHealth) technology and culturally- and linguistically-tailored interpersonal support to increase healthcare engagement of LEP Latino parents and to enable participants to overcome barriers to effective healthcare access and use. Investigators hypothesize that this intervention will measurably increase parent healthcare engagement and that this will positively impact healthcare utilization, quality and the patient/family experience. Increasing healthcare engagement of LEP Latino families and demonstrating positive healthcare impact through a tailored, scalable intervention would create a foundation for larger-scale impact on healthcare disparities for Latino children and a model for increasing engagement of other vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or legal guardian of a singleton US-born infant ≤ 2 months of age
2. Parent or legal guardian age 18 or older
3. Parent or legal guardian self-identified as Latino/a
4. Parent or legal guardian foreign-born
5. Parental report of Spanish as their preferred healthcare language
6. Plan to select Medicaid/Priority Partners insurance for their child with the Johns Hopkins Bayview Medical Center Children's Medical Practice as the primary care site
7. Have a working cellular phone with text message capability and parent reports prior use of text messaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Up to Date Well Child Care | 24 months
  Composite variable of % of AAP recommended well visits completed at intervals 12 and 24 months of age, up to date immunizations and screening at 12 and 24 months
Emergency/Urgent Care Utilization | 24 months
  # of ED/Urgent care visits
Parent experience of care | 12 months
  Use of standard measure of healthcare experiences (Child-CAHPS)

SECONDARY OUTCOMES:
Parent activation | 12 months
Proportion of visits in the the past 12 months with the primary provider | 12 months
Food stamp enrollment | 12 months
Continuous health insurance for the child each of the last 12 months | 12 months
Use of clinic support programs | 12 months

OTHER OUTCOMES:
Intervention delivery | 12 months
  Measurement of intervention activities delivered per participant in the intervention arm
Intervention satisfaction | 12 months
  Quantitative and qualitative measurement of intervention experience for participants in the intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R DeCamp, MD, MSPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roseman D, Osborne-Stafsnes J, Amy CH, Boslaugh S, Slate-Miller K. Early lessons from four 'aligning forces for quality' communities bolster the case for patient-centered care. Health Aff (Millwood). 2013 Feb;32(2):232-41. doi: 10.1377/hlthaff.2012.1085. PMID 23381515
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Derived] Reuland CJ, Godage SK, Wu L, Valenzuela-Araujo D, Cortez JD, Polk S, DeCamp LR. Information and Communication Technology Access and Use Among Low-Income Latino Immigrant Parents. Matern Child Health J. 2021 Dec;25(12):1807-1813. doi: 10.1007/s10995-021-03265-6. Epub 2021 Oct 23. PMID 34687401
- [Derived] DeCamp LR, Godage SK, Valenzuela Araujo D, Dominguez Cortez J, Wu L, Psoter KJ, Quintanilla K, Rivera Rodriguez T, Polk S. A Texting Intervention in Latino Families to Reduce ED Use: A Randomized Trial. Pediatrics. 2020 Jan;145(1):e20191405. doi: 10.1542/peds.2019-1405. PMID 31879276